CLINICAL TRIAL: NCT06262802
Title: In Patients With Large Cystic Lesion Does Volume Reduction Occurs Faster by Using Active Decompression and Distraction Sugosteogenesis Than Using Passive Decompression
Brief Title: Volumetric Changes in Large Cystic Lesions Using Active Decompression and Distraction Sugosteogenesis vs Passive Decompression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radwa Hydar Ragab (Other)
Responsible Party: Sponsor-Investigator, Radwa Hydar Ragab, Principle investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 123123
Record Dates: First submitted 2024-02-07; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Odontogenic Cysts
MeSH Terms: conditions — Odontogenic Cysts

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Device: Active decompression
- Control (Active Comparator)
  Interventions: Device: Active decompression

INTERVENTIONS:
Device: Active decompression — Intracystic active negative pressure

SUMMARY:
Null hypothesis active decompression and distraction sugosteogenesis is not faster than passive decompression in volume reduction of large cystic lesions

ELIGIBILITY:
Inclusion Criteria:

* any patient with large cystic lesion

Exclusion Criteria:

* any patient can't follow home instructions

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Volume change | 2weeks/one and 6 months
  Percentage of volume changes over time